CLINICAL TRIAL: NCT04637620
Title: NMDA Modulation in Major Depressive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH103-REC2-130
Record Dates: First submitted 2020-10-11; First posted 2020-11-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; NMDA; Selective serotonin reuptake inhibitor
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NMDAE (Experimental): An NMDA enhancer
  Interventions: Drug: NMDAE
- SSRI (Active Comparator): Sertraline (selective serotonin reuptake inhibitor)
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Cap

INTERVENTIONS:
Drug: NMDAE — Use of an NMDA enhancer for the treatment of MDD
  Arms: NMDAE
Drug: Sertraline — Use of SSRI as an active comparator
  Arms: SSRI
Drug: Placebo Cap — Use of placebo as a comparator
  Arms: Placebo

SUMMARY:
Most of the current antidepressants for major depressive disorder (MDD) are based upon the monoamine hypothesis which cannot fully explain the etiology of depression. NMDA hypofunction has been implicated in the pathophysiology of depression. Therefore, this study will examine the efficacy and safety as well as cognitive function improvement of an NMDA enhancer (NMDAE) in the treatment of MDD in the adults.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a complex and multi-factorial disorder. Most of the current antidepressants are based upon the monoamine hypothesis which cannot fully explain the etiology of depression. Many patients have significant side effects after treatment with antidepressants which hamper the motivation for treatment and medication adherence. NMDA hypofunction has been implicated in the pathophysiology of depression. MDD is often associated with cognitive deficits which are not necessarily recovered by current antidepressants. The NMDA receptor regulates synaptic plasticity, memory, and cognition. In our previous studies, cognitive improvement has been observed with treatment of NMDA enhancers. Therefore, this study will examine the efficacy and safety as well as cognitive function improvement of NMDAE in the treatment of MDD in the general adults by comparing with sertraline (a selective serotonin reuptake inhibitor [SSRI]) and placebo. The investigators will enroll non-elderly adult patients with MDD for an 8-week treatment. All patients will be randomly assigned into three groups: NMDAE, sertraline, or placebo. The investigators will biweekly measure clinical performances and side effects. Cognitive functions will be assessed at baseline and at endpoint of treatment by a battery of tests. The efficacy of three groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-5 (American Psychiatric Association) diagnosis of MDD
* 17-item Hamilton Rating Scale for Depression total score ≥ 18
* Free of antidepressant drugs for at least 2 weeks
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* Current substance abuse or history of substance dependence in the past 6 months
* History of epilepsy, head trauma, stroke or other serious medical or neurological illness which may interfere with the study
* Bipolar depression, schizophrenia or other psychotic disorder
* Moderate-severe suicidal risks
* Severe cognitive impairment
* Initiating or stopping formal psychotherapy within six weeks prior to enrollment
* A history of severe adverse reaction to SSRIs
* A treatment-resistant history (that is, they have failed to respond to two or more different classes of antidepressants with adequate dosage and treatment duration
* A history of previously received electroconvulsive therapy
* Inability to follow protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Rating Scale for Depression | week 0, 2, 4, 6, 8
  Assessment of depressive symptoms Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.
Change in Global Assessment of Functioning | Week 0, 2, 4, 6, 8
  Assessment of global improvement. Minimum value: 1, maximum value:100, the higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change in Perceived Stress Scale | week 0, 2, 4, 6, 8
  Assessment of stress and anxiety symptoms Minimum value: 0, maximum value:56, the higher scores mean a worse outcome.
Visual Analogue Scale (VAS) | week 0, 2, 4, 6, 8
  Assessment of pain Minimum value: 0, maximum value:10, the higher scores mean a worse outcome.
Clinical Global Impression | week 0, 2, 4, 6, 8
Quality of life (SF-36) | week 0, 8
Visual Continuous Performance Test | week 0, 8
  Assessment of sustained attention
Wisconsin Card Sorting Test | week 0, 8
  Assessment of abstract and shift set
Logical Memory Test of the Wechsler Memory Scale | week 0, 8
  Assessment of episodic memory
Digit Span | week 0, 8
  Assessment of verbal working memory
Spatial Span | week 0, 8
  Assessment of nonverbal working memory
Category Fluency | week 0, 8
  Assessment of speed of processing
Trail Marking A | week 0, 8
  Assessment of speed of processing
WAIS-III Digit Symbol-Coding | week 0, 8
  Assessment of speed of processing
Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) V2.0 | week 0, 8
  Assessment of social cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan